CLINICAL TRIAL: NCT05335811
Title: First-in-Human Assessment of Safety, Biodistribution and Pharmacokinetics of 18F-Fluoro-1-Naphthol (18F-4FN) for PET Imaging
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0784; NCI-2022-01722 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-02-18; First posted 2022-04-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Endocrine Neoplasia
MeSH Terms: conditions — Endocrine Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 4-[18F]Fluoro-1-Naphthol (Experimental): Participants will receive 1 injection of [18F]4FN
  Interventions: Drug: 4-[18F]Fluoro-1-Naphthol

INTERVENTIONS:
Drug: 4-[18F]Fluoro-1-Naphthol — By vein (IV)
  Other Names: [18F]4FN

SUMMARY:
18F-4FN represents a novel PET agent for imaging inflammation. Acute inflammatory signaling through the TLR axis recruits neutrophils and macrophages to inflammatory sites. Both cells activate the production of high energy reactive oxygen species/reactive nitrogen species (RONS), setting off a cascade that can be leveraged to detect the presence of these inflammatory cells by molecular imaging. 18F-4FN is efficiently oxidized by high energy RONS, leading to retention and accumulation in human neutrophil-like cells in vitro, and at the sites of acute inflammation in vivo. Like 18F-FDG, 18F-4FN clears rapidly through the kidney at 1 hr following i.v. injection

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

The primary objective of this first-in-human (FIH) study is to determine the safety, biodistribution, and dosimetry profile of a novel positron emission tomography (PET) imaging tracer, 4-[18F]fluoro-1-naphthol ([18F]4FN), which specifically targets reactive oxygen species (ROS). A currently proposed indication for this radiopharmaceutical (RP) is to non-invasively quantify inflammation by PET/CT imaging.

Exploratory Objectives:

One exploratory objective is to identify preliminary efficacy signals from PET/CT images indicating that the new radiopharmaceutical localized to known or clinically-suspected tissues or regions of inflammation mediated by innate immune-related adverse events (irAE). Another exploratory objective is to determine if a time point other than one-hour post injection will yield clinically meaningful improvements to imaging data.

ELIGIBILITY:
Inclusion Criteria:

* Patient >/= 18 years of age.
* Patients with histologic diagnosis of solid or liquid tumor treated by ICI with evidence of or clinical suspicion of irAE or patients with suspected inflammation.
* Normal range standard renal and liver function tests for age:

eGFR >= 60 mL/min/1.73 m2

Adequate liver function:

Bilirubin ≤ the upper limit of normal (ULN) Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ the ULN

Exclusion Criteria:

* Pregnant or lactating women: pregnant women are excluded from this study because the effects of [18F]4FN in pregnancy are not known. Urine or serum pregnancy test (female </= 60 years of age or childbearing potential) within 24 hours of the PET scan.
* Subjects with contraindications to the use of [18F]4FN including confirmed allergy.
* Patients with a body weight of 400 pounds or more, or a BMI which precludes their entry into the bore of the PET/CT scanner, because the hardware is not intended to support that weight.
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the physician may significantly interfere with study compliance.
* Children below the age of 18 are excluded because of the unknown but potential risk of administration of radiopharmaceuticals to minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To identify preliminary efficacy signals from PET images that correlate with clinical foci of ICI-related irAE. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit Tewari, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05335811/ICF_000.pdf